CLINICAL TRIAL: NCT05448040
Title: Clinical and Histological Assessment of Free Gingival Graft or Collagen Matrix for Socket Sealing After Bone Grafting: a Randomized Controlled Clinical Trial
Brief Title: Clinical and Histological Assessment of Free Gingival Graft or Collagen Matrix for Socket Sealing After Bone Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Salgado de Oliveira (Other)
Responsible Party: Principal Investigator, Gustavo Fernandes, DDS, MSc, PhD, Clinical Lecturer, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 370723 14.4.0000.5374
Record Dates: First submitted 2022-06-24; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Socket Sealing; Free Gingival Graft; Collagen Membrane
Keywords: Alveolar sealing; Free gingival graft; Autogenous graft; Collagen matrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen (Experimental): This group received a bone graft (xenograft) and had the socket covered with a collagen membrane, in order to protect the bone graft inserted and seal the socket.
  Interventions: Procedure: Socket preservation
- Free gingival graft (Experimental): This group received a bone graft (xenograft) biomaterial and had the socket covered with a free gingival graft material, in order to protect the bone graft inserted and seal the socket.
  Interventions: Procedure: Socket preservation

INTERVENTIONS:
Procedure: Socket preservation — Tooth extraction and preservation with a biomaterial

SUMMARY:
The goal of this study was to compare, clinical and histologically, the use of the suine collagen matrix (Mucograft Seal [MS], Geisthlich®) and the free gingival graft (FGG) for the alveolar sealing after inserted bone graft biomaterial. It was included 18 patients with tooth referred to extraction (maxilar incisives, canines, or pre-molars) which were randomly divided in 2 groups, according to the material for alveolus sealing: control (FGG) and test (MS). After the minimally traumatic extraction, all the alveoli were filled with bovine mineral matrix (Bio-Oss®), and the material for alveolar sealing were positioned and stabilized with sutures. The follow-up (clinical and photographic) happened on the immediate post-operatory period, and with 3, 7, 15, 30, 60, 90, and 120 days. After 120 days, before implant placement, tissues samples were obtained with a 3.5mm punch scalpel for histological analysis. Qualitative information related to the patient's perception considering the treatment were collected.

ELIGIBILITY:
Inclusion criteria

* patients ASA I
* patients requiring single tooth extraction in the site between #4 to #13
* patients without enough bone volume for immediate implant placement.

Exclusion criteria

* patients with general contraindications for implant surgery
* pregnant or lactating women
* patients with untreated periodontitis
* bruxism or severe clenching
* immunosuppressed
* patients with a previous history of irradiation of the head and neck area
* uncontrolled diabetes
* heavy smoker (>10 cigarettes/day)
* poor oral hygiene and low motivation
* use of bisphosphonates
* substance abuse such as alcohol or drugs and psychiatric disorders.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Radiographic and clinical analysis | 6 months
  Socket preservation with xenograft biomaterial and another one to seal it (FGG or collagen membrane).
  Radiographic analysis - PA (periapical x-rays) comparing groups and periods of the follow-up. It was performed descriptive comparative analysis.
  Clinical evaluation - bleeding on probing (dichotomic analysis), ISQ (torque achieved - Osstell), qualitative analysis (questionnaire with 8 questions), and subjective appraisal of the soft tissue healing (according to the period of evaluation).

SECONDARY OUTCOMES:
Histological analysis - Gingiva | 6 months
  Gingival thickness obtained from the local tissue was evaluated through histological analysis (optical binocular microscope); assessment of the epithelial and connective layers (micrometers).

CONTACTS AND LOCATIONS:
Overall Officials: Joly, PhD, Principal Investigator — Sao Leopoldo Mandic
Locations (1):
- UM - POM Dpt, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No.